CLINICAL TRIAL: NCT06575673
Title: Effect of an Internet-based Dialectical Behaviour Therapy-informed Skills Training for Promoting Smoking Cessation and Improving Psychological Distress of Smokers: A Pilot Randomised Controlled Trial
Brief Title: An Internet-based Dialectical Behaviour Therapy-informed Skills Training for Promoting Smoking Cessation and Improving Psychological Distress of Adult Smokers.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ho Long Kwan, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07210048
Record Dates: First submitted 2024-08-19; First posted 2024-08-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Smoking
Keywords: Dialectical behaviour therapy; Skills training; Internet-based intervention; Psychological distress; Adult smokers; Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DBT-ST group (Experimental): Participants in the intervention group will receive the DBT-ST by means of a free video-communication app. Over the next 14 weeks from the baseline, participants will receive two individual sessions (30-45 mins) and 12 group therapy sessions (120-minute)
  Interventions: Behavioral: Internet-based dialectical behaviour therapy-informed skills training
- TAU (Other): Participants in the control group will receive a smoking cessation booklet published by the Hong Kong Council on Smoking and Health that provided information on the negative health consequences of smoking, reasons to quit, strategies for quitting, smoking cessation services available in Hong Kong, and a public Quitline number (usual care). Participants will also receive a monthly health education for three months that provides general health information and sharing sessions, which is one of the routine care for smokers during the first 3-4 months after they seek help for smoking problem (waiting period for further intervention).
  Interventions: Behavioral: Monthly health education

INTERVENTIONS:
Behavioral: Internet-based dialectical behaviour therapy-informed skills training — Adaptive applications of DBT-ST for smokers with psychological distress
  Arms: DBT-ST group
Behavioral: Monthly health education — General health information and sharing sessions
  Arms: TAU

SUMMARY:
1. To determine the feasibility, acceptability, and preliminary effects of an internet-based DBT-ST for promoting smoking abstinence/reduction and improving psychological distress/emotional regulation in adult smokers
2. To explore the participants' experiences and perceptions (e.g., perceived benefits/weaknesses) towards the proposed intervention

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese aged 18-64 years
* Had smoked at least one cigarette per day over the previous three months
* Indicate psychological distress as measured by the Depression, Anxiety, and Stress Scale-21
* Have an intention to stop smoking
* Have an electronic device and are willing to receive interventions via the internet

Exclusion Criteria:

* Experiencing psychotic disorders/cognitive impairment/communication problems
* Participating in other smoking cessation programs or related psychosocial interventions

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated 7-day PPA (an exhaled CO test and a salivary cotinine test) | Baseline, 3-month post-intervention
  Participants who self-reported not smoking within the past seven days will be invited to attend a biochemical verification test of smoking abstinence
Level of psychological distress | Baseline, 3-month post-intervention
  Symptoms of depression, anxiety and stress measured by the Chinese version of Depression, Anxiety, and Stress Scale-21

SECONDARY OUTCOMES:
Self-reported 7-day PPA | Baseline, 3-month post-intervention
  Self-reporting of complete abstinence for at least seven days prior to assessment
Self-reported smoking reduction of at least 50% | 3-month post-intervention
  Participants will report the number of cigarette they consume and the number will be compared to the number at baseline
Quit attempts | Baseline, 3-month post-intervention
  The number of times that the participant engage in a period of intentional abstinence of more than 24 hours in the previous three months
Emotion dysregulation | Baseline, 3-month post-intervention
  Levels of emotion dysregulation measured by the Chinese version of the Difficulties in Emotion Regulation Scale (DERS)
Distress tolerance | Baseline, 3-month post-intervention
  Perceived ability to tolerate emotional distress measured by the Chinese version of the Distress Tolerance Scale (DTS)

OTHER OUTCOMES:
Acceptability | 3-month post-intervention
  Client Satisfaction measured by the 8-item Client Satisfaction Questionnaire-8
Feasibility of the intervention | 3-month post-intervention
  Recruitment rate
Feasibility of the intervention | 3-month post-intervention
  Intervention engagement in terms of time spent on each session and participation rates
Feasibility of the intervention | 3-month post-intervention
  Attrition rates
Semi-structured interview | 3-month post-intervention
  Individual semi-structured interviews will be conducted at post-intervention to explore participants' experiences/perceptions of the internet-based DBT-ST, as well as their comments on the appropriateness/comprehensiveness of the content/frequency of the intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Hospital Authority, Tai Po, New Territories
  - Hospital Authority, Hong Kong